CLINICAL TRIAL: NCT04373122
Title: CPR-REBOA: Improving Outcome of Prehospital Cardiopulmonary Resuscitation With Balloon Occlusion of the Descending Aorta
Brief Title: REBOA in Out-of-hospital Cardiac Arrest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: City of Bern (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-02039
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Out-of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- REBOA (Experimental): Insertion of the ER-REBOA Catheter during ongoing CPR
  Interventions: Device: REBOA

INTERVENTIONS:
Device: REBOA — Resuscitative Endovascular Balloon Occlusion of the Aorta

SUMMARY:
Unexpected cardiac arrest is a frequent and devastating event with a high mortality and morbidity. Half of the patients who survive to ICU admission ultimately die because of hypoxic-ischemic encephalopathy. With CPR and advanced life support, blood and oxygen delivery to heart and brain is preserved until circulation is restored. During CPR, coronary perfusion pressure is a significant predictor of increased rates of return of spontaneous circulation (ROSC) and survival to hospital discharge, while cerebral perfusion pressure is crucial for good neurologic outcome. Existing efforts to reduce mortality and morbidity focus on rapid recognition of cardiac arrest, initiation of basic and advanced life support (ALS), and optimization of post-arrest care.

Clamping the descending aorta during cardio-pulmonary resuscitation (CPR) should redistribute the blood flow towards brain and heart. Animal models of continuous balloon occlusion of the aorta in non-traumatic cardiac arrest have shown meaningful increases in coronary artery blood flow, coronary artery perfusion pressure and carotid blood flow, leading to improved rates of ROSC, 48h-survival and neurological function.

In humans, occlusion of the aorta using a REBOA catheter in the management of non-compressible abdominal or pelvic hemorrhage has shown improvements in hemodynamic profiles and has proved to be feasible in both, clinical and preclinical settings for trauma patients in hemorrhagic shock. These promising data provide an opportunity to improve outcome after cardiac arrest in humans too. The investigators have developed a protocol for the reliable and safe placement of a REBOA-catheter during cardiac arrest in a clinical setting (see ClinicalTrials.gov Identifier: NCT03664557).

Damage to heart and brain from lack of oxygen supply occurs during the first minutes following cardiac arrest. It is therefore crucial to apply any measure to improve efficacy of CPR early in the course of events and therapy. After proving feasibility in a clinical setting in the trial mentioned above, the next logical step and specific goal of this study is to transfer this protocol to the preclinical setting, and to investigate the effect of temporary endovascular occlusion of the descending aorta on the efficacy of CPR early in the course of treatment of out-of hospital cardiac arrest by means of an increase in blood pressure.

DETAILED DESCRIPTION:
Unexpected cardiac arrest is a devastating event with a high mortality and morbidity. Half of the patients who survive to ICU admission ultimately die because of hypoxic-ischemic encephalopathy (HIE). As outcome after cardiac arrest is depending on time and amount of oxygen delivery to heart and brain, preserving myocardial and cerebral perfusion in the event of cardiac arrest by the means of effective cardio-pulmonary resuscitation (CPR) is of utmost importance. During CPR Coronary perfusion pressure is a significant predictor of increased rates of return of spontaneous circulation (ROSC) and survival to hospital discharge, while cerebral perfusion pressure is crucial for good neurologic outcome. The absence of ROSC despite prolonged high quality and efficient initial basic life support (BLS) followed by traditional ALS ends finally in neuronal damage and death.

For those patients not qualifying for eCPR or in areas where this highly invasive approach is not readily available, existing efforts to reduce mortality and morbidity focus on rapid recognition of cardiac arrest, initiation of basic and advanced life support (ALS), and optimization of post-arrest care.

Clamping the descending aorta during cardio-pulmonary resuscitation (CPR) should redistribute the blood flow towards brain and heart. Animal models of continuous balloon occlusion of the aorta in non-traumatic cardiac arrest have shown meaningful increases in coronary artery blood flow, coronary artery perfusion pressure and carotid blood flow, leading to improved rates of ROSC, 48h-survival and neurological function.

In humans, occlusion of the aorta using a REBOA catheter in the management of non-compressible abdominal or pelvic hemorrhage has shown improvements in hemodynamic profiles and has proved to be feasible in both, clinical and preclinical settings for trauma patients in hemorrhagic shock. These promising data provide an opportunity to improve outcome after cardiac arrest in humans too. For an ongoing study evaluating its feasibility, the investigators have developed a protocol for the reliable and safe placement of a REBOA-catheter during cardiac arrest in a clinical setting (see ClinicalTrials.gov Identifier: NCT03664557).

Damage to heart and brain from lack of oxygen supply occurs during the first minutes following cardiac arrest. It is therefore crucial to apply any measure to improve efficacy of CPR early in the course of events and therapy. After proving feasibility in a clinical setting in the trial mentioned above, the next logical step and specific goal of this study is to transfer this protocol to the preclinical setting, and to investigate the effect of temporary endovascular occlusion of the descending aorta on the efficacy of CPR early in the course of treatment of out-of hospital cardiac arrest by means of an increase in blood pressure.

The objectives are to investigate the effect of resuscitative endovascular balloon occlusion of the descending aorta early in the course of cardiac arrest therapy on blood pressure, cerebral oxygenation and endtidalCO2- Data collection allowing for sample calculation for a large outcome study

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from refractory Out-of-hospital cardiac arrest (OHCA) of presumed cardiac origin, defined as failure to achieve stable ROSC within 10 min of fully established standard care (ALS) which do not qualify for extracorporeal cardiac life support (e-CPR).
* Witnessed Arrest
* Interval from collapse to initiation of sufficient (lay) CPR less than 5 minutes

Exclusion Criteria:

* Patients whose underlying disease limit survival and resuscitation measures are stopped after initial assessment, or evaluation reveals futile clinical situation
* Patients with advanced directives or living will which excludes CPR
* Age < 18 years (device certified >18 years)
* Qualifying for other treatment options, namely eCPR (CPR with extracorporeal membrane oxygenation (ECMO) as life assist device)
* Unwitnessed arrest with asystole as first documented rhythm
* etCO2 below 15mmHg
* Patients in whom no femoral arterial access site cannot accommodate a 7 Fr (minimum) introducer sheath
* Known to have an aortic diameter larger than 32 mm
* Evidence or suspicion of thoracic trauma
* Inability to guarantee standard ALS measures during performance of the REBOA maneuver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of blood pressure | 10 minutes
  Increase of blood pressure after balloon occlusion of the aorta

SECONDARY OUTCOMES:
Change of NIRS | 10 minutes
  Increase of NIRS (near-infrared reflectance spectroscopy) after balloon occlusion of the aorta
Change of etCO2 | 10 minutes
  Increase of etCO2 (end-tidal CO2) after balloon occlusion of the aorta

OTHER OUTCOMES:
Outcomes | up to 6 months
  Neurological Outcomes measured by CPC

CONTACTS AND LOCATIONS:
Overall Officials: Anja Levis, MD, Principal Investigator — University of Bern, Inselspital
Locations (1):
- Departement of Intensive Care Medicine - University Hospital Bern - Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual request